CLINICAL TRIAL: NCT03382704
Title: Vellus Hair Loss as a Marker for Peri-ocular Malignancy
Status: Withdrawn | Type: Observational
Why Stopped: withdrawn prior to approvals being given
Sponsor: NHS Lothian (Other Government)
Collaborators: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 229755
Record Dates: First submitted 2017-12-13; First posted 2017-12-26 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-09

CONDITIONS: Skin Cancer Face
Keywords: Peri-ocular
MeSH Terms: interventions — Physical Examination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Pathology samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing biopsy: Patients undergoing biopsy (incisional or excisional) of peri-ocular lesions. Pre-operative examination for presence or absence of vellus hairs
  Interventions: Diagnostic Test: Examination for presence or absence of vellus hairs

INTERVENTIONS:
Diagnostic Test: Examination for presence or absence of vellus hairs — Pre-operative examination for presence or absence of vellus hairs

SUMMARY:
Skin cancers around the eye are common, but so are other lid lumps. It is useful to be able to tell which lumps are likely to be cancer.

This study looks at whether the loss of fine hairs (vellus hairs) on the skin are a good indicator of whether a lump is a skin cancer or not.

The investigators are recruiting patients who have lid lumps who haven't had a biopsy before, who would be having a biopsy as part of their treatment, and seeing whether those who have loss of the fine skin hairs are the same as those who have skin cancer confirmed on their biopsy.

The study doesn't involve any extra examinations or treatments for participants. The investigators look at the patients before the biopsy as part of their usual care, and take a note of whether or not they have lost the fine hairs at this stage.

The main benefit of participating is that the medical community has better evidence about which lid lumps are likely to represent skin cancer, helping future diagnosis.

There are no additional risks to participating. The risks of biopsy are unchanged whether patients participate in the study or not.

The study is run from the Princess Alexandra Eye Pavilion in Edinburgh.

The investigators aim to start the study in Spring 2020, and will most likely recruit for 6 months depending on the number of participants recruited.

There is no additional funding from any source at present - the work will be undertaken by doctors in their research time.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing biopsy for peri-ocular lesion

Exclusion Criteria:

* Age under 18; previous biopsy or excision on the same lid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All cases undergoing incision or excision biopsy of peri-ocular lesions at the study institution during the study period
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Vellus hair presence/absence | Day 1
  Examination for the presence or absence of vellus hairs prior to biopsy
Biopsy result | On receipt of biopsy result from pathology lab (~1 week)
  Biopsy result looking for malignancy

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Peden, MA; MBBS; FRCOphth, Principal Investigator — NHS Lothian
Locations (1):
- Princess Alexandra Eye Pavilion, Edinburgh, Midlothian, United Kingdom

IPD SHARING:
Plan to Share IPD: No